CLINICAL TRIAL: NCT07011160
Title: Neural Substrates Underlying Adaptations in Manual Dexterity of Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Roger Enoka, PI, University of Colorado, Boulder
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 1R01NS141829-01A1
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Aging Hands
Keywords: manual dexterity; force steadiness; motor units; neuroplasticity
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pegboard time (Experimental): Participants will be assigned to a group of slow or fast improvers based on the decrease in pegboard time after an initial familiarization session.
  Interventions: Behavioral: Familiarization
- Force-steadiness practice (Experimental): Participants will complete three training sessions in which they perform force-steadiness tasks either alone (sham) or paired with transcutaneous electrical nerve stimulation (TENS). One-half of the participants in each improver group will be to each of these practice groups.
  Interventions: Behavioral: Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Behavioral: Transcutaneous electrical nerve stimulation (TENS) — Force-steadiness training will be performance either without (sham) or paired with TENS.
  Arms: Force-steadiness practice
Behavioral: Familiarization — Participants will perform 25 trials of the Grooved Pegboard Test
  Arms: Pegboard time

SUMMARY:
Age-related declines in motor function can compromise independence and quality of life. This project examines how practice and somatosensory stimulation reshape the neural control of hand muscles in older adults, leveraging neuroplasticity to enhance dexterity. By identifying modifiable neural mechanisms that underlie improved motor performance, this research lays the groundwork for targeted, non-invasive interventions that can be translated into clinical and community settings to support healthy aging and functional independence.

DETAILED DESCRIPTION:
Managing fine motor function is essential for independence and quality of life in older adults. However, the neural mechanisms underlying age-related declines in manual dexterity remain poorly understood. Traditional models of motor control suggest that the nervous system coordinates movement through shared motor commands across muscles-so-called "motor modules" or "muscle synergies". Yet, emerging evidence reveals that synaptic inputs to motor neurons can vary even within a single muscle, challenging this muscle-level concept and prompting a shift toward more a granular, motor-unit level framework. These "motor unit modes" offer a more accurate representation of the neural architecture of motor control.

This project will be the first to investigate whether improvements in manual dexterity-a core marker of neurological health in aging-are associated with neuroplastic changes in the strength of functionally relevant motor unit modes. Older adults (54-89 yrs) will practice a test of manual dexterity (Grooved Pegboard) with or without performance-enhancing transcutaneous electrical nerve stimulation (TENS). Outcomes will include force steadiness and motor unit activity derived from high-density electromyography during low-intensity contractions.

Our central hypothesis is that improvements in manual dexterity will be mediated by neuroplastic strengthening of functionally relevant motor unit modes. The project has three specific aims:

1. Characterize short-term neuroplastic adaptations following task familiarization.
2. Determine the effects of steady-contraction training on neuromuscular control.
3. Evaluate the added benefit of somatosensory augmentation with TENS.

Innovation. This study introduces two key innovations: (1) It quantifies, for the first time, the extent to which improvements in a dynamic behavior are mediated by changes in shared synaptic inputs across motor units during low-intensity contractions; (2) it evaluates the capacity of TENS-induced somatosensory feedback to boost neuroplasticity in the aging motor system.

Expected Outcomes. We expect that gains in force steadiness and pegboard performance will strongly correlate with increased strength and consistency of motor unit modes. These findings will clarify the neural mechanisms underlying motor adaptation in older adults and define new markers for assessing motor function.

Impact. Aligned with the goals of PA-25-303 and the missions of NINDS and NIA, this research will generate foundational knowledge of spinal motor control and establish motor unit modes as a new biomarker for evaluating motor function and therapeutic efficacy. This work has the potential to inform targeted interventions aimed at preserving dexterity and independence in older individuals and those with neurological dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Community-dwelling men and women who are 54-89 years of age and able to give fully informed consent; able to read, write, and speak English to ensure safe participation in the project; and able to arrange own transportation to Boulder campus.

Exclusion Criteria:

Cognitive impairment, major psychiatric condition, or unstable depressive disorder that would influence the ability to understand the study and cooperate fully in the proposed protocols; any progressive neurological, muscular, cardiovascular, or skeletal disorder that limits participation, such as (but not limited to) (1) amyotrophic lateral sclerosis, multiple sclerosis, multiple system atrophy, muscular dystrophy, myasthenia gravis, Parkinson's disease, spinal muscular atrophy, spinocerebellar ataxia, or spasticity; (2) congenital, mitochondrial, or thyrotoxic myopathies, fibromyalgia, or myositis; (3) peripheral neuropathy, diabetes, or hypertension; or (4) cancer, gout, osteoarthritis with severe pain, or rheumatoid arthritis; chronic pain condition that would impair the ability to participate in the study; currently taking prescribed medication known to influence neuromuscular function, such as carisoprodol, cyclobenzaprine, metaxalone, and methocarbamol; function-limiting injury to the hands, arms, shoulders, neck, or legs; recent hospitalization (within the last 3 months) or enforced bedrest/sedentary state; inability to attend the evaluation and practice sessions in 2 weeks.

Ages: 54 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-03-30 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
Grooved Pegboard Test | From enrollment until the end of the study at 2 weeks.
  Time taken to insert 25 keyhole-shaped pegs into matching holes on the pegboard.
Force steadiness | From enrollment until the end of the study at 2 weeks.
  Coefficient of variation for force during low-intensity isometric contractions.
Motor unit modes | From enrollment until study completion at 2 weeks.
  The subsets of motor units in hand-forearm muscles that exhibit correlated modulation of discharge rate during low-intensity isometric contractions. The motor unit activity will be identified from high-density surface electromyography with grid electrodes.

CONTACTS AND LOCATIONS:
Overall Officials: Roger M Enoka, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
In this proposed project, the cleaned, item-level spreadsheet data for all variables will be shared openly, along with example quantifications and transformations from initial raw data. Final files used to generate specific analyses to answer the Specific Aims and related results will also be shared. The rationale for sharing only cleaned data is to foster ease of data reuse.

REFERENCES:
- [Background] Tvrdy T, Henry M, Enoka RM. Influence of the variability in motor unit discharge times and neural drive on force steadiness during submaximal contractions with a hand muscle. J Neurophysiol. 2025 Feb 1;133(2):697-708. doi: 10.1152/jn.00333.2024. Epub 2025 Jan 17. PMID 39823197
- [Background] Daneshgar S, Tvrdy T, Enoka RM. Explaining the influence of practice on the grooved pegboard times of older adults: role of force steadiness. Exp Brain Res. 2024 Aug;242(8):1971-1982. doi: 10.1007/s00221-024-06878-9. Epub 2024 Jun 25. PMID 38916760
- [Background] Daneshgar S, Tvrdy T, Enoka RM. Practice-Induced Changes in Manual Dexterity of Older Adults Depend on Initial Pegboard Time. Med Sci Sports Exerc. 2023 Nov 1;55(11):2045-2052. doi: 10.1249/MSS.0000000000003245. Epub 2023 Jun 27. PMID 37379250